CLINICAL TRIAL: NCT05314608
Title: Prospective Study of Bone Pathologies Resulting From Acute or Chronic Injury Treated With IntraOsseous BioPlasty® (IOBP®) Surgical Technique
Brief Title: Knee Related Subchondral Bone Lesions Treated With IOBP
Acronym: IOBP
Status: Recruiting | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20085
Record Dates: First submitted 2022-02-23; First posted 2022-04-06 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Subchondral Cyst
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with subchondral bone pathology: Subjects with subchondral bone pathology
  Interventions: Combination Product: IntraOsseous BioPlasty® (IOBP®) Surgical Technique into the knee

INTERVENTIONS:
Combination Product: IntraOsseous BioPlasty® (IOBP®) Surgical Technique into the knee — Injection of a biologic mixture (BMC and allograft) into the subchondral bone lesion

SUMMARY:
The study will be a prospective, multicenter clinical study evaluating clinical and patient reported outcome measures of subjects receiving IOBP® surgical technique using Angel cPRP and BMA processing system to treat subchondral bone pathology (SBP).

DETAILED DESCRIPTION:
The study will be a prospective, multicenter, clinical study, enrolling both male and female patients. Subjects will be identified among the investigators' patient population scheduled for the IOBP® procedure and as being diagnosed with symptomatic SBP that have failed conservative management. IRB approval will be obtained by each participating institution.

The primary outcome measure is adverse event evaluation to determine whether IOBP® can prevent further surgical intervention (i.e., knee replacement surgery, HTO, or calcium phosphate stabilization of SBP) when used to treat symptomatic SBP of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, sign and complete informed consent
2. Male or female subject between the ages of 18-60 years
3. Subject has had pain for greater than three months
4. Subjects with single SBP in tibia or femur confirmed by minimum 1.5T MRI (including coronal, axial, sagittal, lateral femur, and lateral tibia views) and are candidates for an IOBP® procedure
5. Subject has stable ligaments
6. Subject has neutral alignment (max 5° varus or valgus)
7. Subject has a VAS score greater than or equal to five
8. Subject is scheduled to undergo surgical intervention using IOBP®

Exclusion Criteria:

1. Subject has diabetes Type I, Type II uncontrolled, or Type II insulin dependent
2. Subject has had lower extremity surgery within six months
3. Subject has had more than two prior surgical procedures in the operative leg
4. Subject has a neuromuscular condition
5. Subject has a current infection
6. Subject has a BMI >35
7. Subject has subchondral bone collapse or Kellgren Lawrence grade IV osteoarthritis
8. Subject has joint surface collapse in late stage avascular necrosis
9. Subject has majority of pain associated with alternate conditions
10. Subject has had subchondral bone pathology caused by acute trauma
11. Subject is not neurologically intact.
12. Subject has history of invasive malignancy (except non-melanoma skin cancer)
13. Subject that has a planned or scheduled additional surgery within the course of the study (lower extremity)
14. Subject has an active substance abuse problem
15. Subject is currently taking narcotic pain medication
16. Subject is pregnant or planning to become pregnant
17. Subject is on worker's compensation
18. Subject has a concomitant procedure not including meniscectomy, synovectomy, chondroplasty, or removal of loose body
19. Inability to complete study requirements and follow-up visits
20. Subject that has a bone marrow aspiration that does not meet 60cc

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be identified among the investigators' patient population scheduled for the IOBP® procedure and as being diagnosed with symptomatic SBP that have failed conservative management.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Prevention of additional surgery into the target knee | 5 years
  To evaluate if IOBP® procedure will prevent further surgical intervention (i.e., knee replacement surgery, HTO, or calcium phosphate stabilization of SBP) when used to treat symptomatic SBP of the knee.

SECONDARY OUTCOMES:
Visual Analog Pain Scale (VAS) | Collected at pre-op, 1 week post-op, 6 weeks post-op, 3 months post-op, 6 months post-op , 1 years post-op , 2 years post-op, 3 years post-op , 4 years post-op and 5 years post-op.
  Patient reported pain scale using a 10 cm scale with a numeric rating of 0 to 10, with 0
International Knee Documentation Committee Subjective Knee Evaluation Form | knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury.
  A patient-oriented questionnaire that assesses symptoms and function in daily living activities. The purpose of this study was to validate the IKDC Subjective Knee Form in a large patient population with various knee disorders.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Collected at pre-op, 1 week post-op, 6 weeks post-op, 3 months post-op, 6 months post-op , 1 years post-op , 2 years post-op, 3 years post-op , 4 years post-op and 5 years post-op
  A knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury.
X-rays of the knee | 6 months and 1 year
  Images include weight-bearing AP, 45 degree weight bearing PA, lateral and merchant views. Images taken to determine location and status of subchondral bone lesion.
MRI of the knee | 6 months and 1 year
  Minimum 1.5 Tesla MRI (including coronal, axial, sagittal, lateral femur, and lateral tibial views). Image taken to determine location and status of subchondral bone lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, Principal Investigator — Andrews Research and Education Foundation
Locations (5):
- United States (5):
  - University of Colorado Sports Medicine, Denver, Colorado
  - Andrews Research and Education Foundation, Gulf Breeze, Florida
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - The Ohio State University, Columbus, Ohio
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No